CLINICAL TRIAL: NCT07192419
Title: Promoting Aging and Thriving With HIV (PATH)-Implementation of a Tailored Geriatric Assessment and Management Strategy for HIV Care Settings
Brief Title: Promoting Aging and Thriving With HIV
Acronym: PATH
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Meredith Greene, Associate Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 27767; K76AG064545-01 (NIH)
Record Dates: First submitted 2025-08-27; First posted 2025-09-25 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: HIV (Human Immunodeficiency Virus); Geriatric; Geriatric Assessment; HIV; HIV - Human Immunodeficiency Virus
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Seroconversion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Usual care participants will receive HIV and aging information before their regular medical appointment.
- PATH (Experimental): The PATH group will undergo an aging assessment using the PATH toolkit before their regular medical appointment.
  Interventions: Behavioral: Promoting Aging and Thriving with HIV (PATH)-Implementation of a Tailored Geriatric Assessment and Management Strategy for HIV Care Settings

INTERVENTIONS:
Behavioral: Promoting Aging and Thriving with HIV (PATH)-Implementation of a Tailored Geriatric Assessment and Management Strategy for HIV Care Settings — For the intervention arm, participants will be sent geriatric assessment questions through the patient portal in advance of a routine HIV appointment. If the participant is unable to complete the questions in advance, they will be done with the help of a research coordinator to go through on the day of appointment. Every attempt will be made to ensure the assessment can be done in advance of the appointment, however the study team will allow for visits after the regular appointment as in which case the provider will receive results after the patient has left clinic.
  The provider will receive the PATH assessment responses and a discussion guide with suggested initial management steps. The provider ultimately determines with the participant when and if they will address concerns identified (that visit or future visit) based on participant priorities. The patient participant will also receive a copy of their screening results.
  Arms: PATH

SUMMARY:
The pilot is an intervention of a geriatric assessment and management tool (PATH) in outpatient HIV clinics.

DETAILED DESCRIPTION:
This will be a Pilot, two-arm, randomized parallel-group, clinical trial with blinded research staff of a Geriatric assessment and management tool vs usual care to evaluate the feasibility, acceptability, and preliminary efficacy of the tool on quality of life for older adults with HIV.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 or older
* Receive HIV care (at least 1 visit at the same site within the past 12 months) from either Eskenazi Health IDC or LifeCare clinics,
* Able to provide informed consent

Exclusion Criteria:

* Patients who are long-term nursing home residents
* Patients who are receiving geriatric care services, however will liberalize this criteria if difficulty with recruitment

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-17 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Feasibility: recruitment and retention | Recruitment day one, throughout the study to final assessment six months post baseline of the last participant.
  Feasibility will be measured by tracking the number of participants approached, enrolled, retained, observations by study team throughout study.
Feasibility: patient/provider experience | After completing final outcomes at the 6 month assessment (or earlier if difficulty with recruitment/retention) patients and providers will be invited to participate in an optional qualitative interview.
  Feasibility will be measured by qualitative Interviews with patients and providers. Interview questions will be used to derive personal anecdotes of the patient/provider experience pertaining to the feasibility of the study.
Acceptability; General attitudes, perception of intervention | After completing final outcomes at the 6 month assessment (or as needed if difficulty with recruitment/retention) patients and providers will be invited to participate in an optional qualitative interview.
  Acceptability will be measured by qualitative Interviews with patients and providers. Interview questions will be used to derive personal anecdotes of the patient/provider general attitudes, perception of intervention.

SECONDARY OUTCOMES:
Impact of PATH Outcomes: measured by identification of geriatric conditions | Geriatric Conditions will be measured through chart review at baseline, 3month, and 6 month assessments to determine overall change from baseline.
  To evaluate the impact of PATH HIV Outcomes the study will look at change from baseline in patient geriatric conditions. This study hypothesizes that compared to usual care, PATH participants will have more geriatric conditions identified and managed as compared to baseline geriatric conditions.
Impact of PATH Outcomes: measured by addressing unmet needs. | Unmet needs will be measured through survey questions and chart review at baseline, 3month, and 6 month assessments.
  Evaluate the impact of PATH HIV on addressing unmet needs of older adults living with HIV. This study hypothesizes that compared to usual care, PATH participants will have more psychosocial needs addressed compared to the number of unmet needs at baseline.
Quality of life as measured by Medical Outcomes 36-Item Short Form Survey (SF-36) | Quality of life will be measures at baseline, 3 months and 6 months post baseline assessments.
  Evaluate the preliminary impact of PATH on health-related quality of life for older adults with HIV using the Medical Outcomes 36-Item Short Form Survey (SF-36). This study hypothesizes that compared to usual care, intervention recipients will have improved quality of life as measured by SF-36. The SF-36 includes eight scales measuring domains of physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. These scores can be combined into a Mental Component Summary Score and a Physical Component Summary Score. Component summary scores range from 0 (poor) to 100 (excellent) with the higher scores representing higher physical/mental health respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Meredith Greene, MD, Principal Investigator — Indiana University School of Medicine, and Regenstrief Institute; IU Center for Aging Research
Locations (2):
- United States (2):
  - Eskenazi Health, Indianapolis, Indiana
  - IU Health LifeCare, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No